CLINICAL TRIAL: NCT05737745
Title: The Initial Efficacy of FitEx for Endometrial Cancer Survivors: A Pilot Randomized Controlled Trial of a Walking Promotion Program With or Without Yoga
Brief Title: FitEx for Endometrial Cancer Survivors: Initial Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Shannon Armbruster, Principal Investigator, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-22-1727; UL1TR003015 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Cancer; Obesity; Sedentary Behavior; Quality of Life; Survivorship
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Sedentary Behavior | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Endometrial cancer survivors will receive standard survivorship care including a one-time educational newsletter about survivorship physical activity and nutrition recommendations. Fitbits will be given to track physical activity.
- FitEx-ECS (Experimental): Endometrial cancer survivors and their support team members (as a group of one survivor and their team) will complete the FitEx-ECS intervention program, with a focus on walking. Fitbits will be given to track physical activity.
  Interventions: Behavioral: Self-monitoring; Behavioral: Group-dynamics; Behavioral: Weekly virtual sessions- Standard; Behavioral: Newsletters- Standard
- FitEx-ECS+ Yoga (Experimental): Endometrial cancer survivors and their support team members (as a group of one survivor and their team) will complete the FitEx-ECS+yoga intervention program, with a focus on postures, breathwork, and mindfulness. Fitbits will be given to track physical activity.
  Interventions: Behavioral: Self-monitoring; Behavioral: Group-dynamics; Behavioral: Newsletters- Yoga; Behavioral: Weekly virtual sessions- Yoga

INTERVENTIONS:
Behavioral: Self-monitoring — Tracking physical activity and fruit/vegetable intake.
  Arms: FitEx-ECS; FitEx-ECS+ Yoga
Behavioral: Group-dynamics — Survivors act as team captains, facilitating interactions between themselves and their support team members and providing goal directed feedback.
  Arms: FitEx-ECS; FitEx-ECS+ Yoga
Behavioral: Weekly virtual sessions- Standard — Weekly 30 minute virtual sessions include support group/team building sessions and 15 minutes of physical activity.
  Arms: FitEx-ECS
Behavioral: Newsletters- Standard — Weekly newsletters support attainment of physical activity and nutrition goals.
  Arms: FitEx-ECS
Behavioral: Newsletters- Yoga — Weekly newsletters support attainment of physical activity and nutrition goals, while including mindfulness principles.
  Arms: FitEx-ECS+ Yoga
Behavioral: Weekly virtual sessions- Yoga — Weekly 30 minute virtual sessions include support group/team building sessions and 15 minutes of yoga.
  Arms: FitEx-ECS+ Yoga

SUMMARY:
The goal of this clinical trial is to compare physical activity outcomes between endometrial cancer survivors randomized to 1 of 3 conditions: 1) usual care, 2) FitEx, 3) FitEx+yoga. Survivors randomized to FitEx groups will recruit ~3 support team members to complete the intervention with them. The main question[s] it aims to answer are:

* Do FitEx groups undertake more physical activity than the usual care group?
* Are there differences in quality of life, self-compassion, flourishing, self-efficacy, social support, habit formation, and fruit /vegetable consumption

Participants will:

* Wear a Fitbit
* Complete surveys
* Participate in 30 minute weekly virtual meetings (FitEx groups only)
* Receive weekly newsletters (FitEx groups only)

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the initial efficacy of FitEx, a physical activity tracking and promotion program, and FitEx+yoga for endometrial cancer survivors (ECS), with focus on improvement of moderate-vigorous physical activity (MVPA) at the completion of the 8-week program. Specifically, this project will recruit early stage ECS with obesity to be randomized to 1 of 3 conditions: 1) usual care, 2) FitEx, 3) FitEx+yoga. ECS in either intervention condition will each select ~3 friends or family members to be their support members (minimum 2 and maximum 5). All ECS will receive a Fitbit to track their MVPA. We will then compare secondary ECS outcome measures between intervention and control groups including quality of life, self-compassion, flourishing, self-efficacy, social support, habit formation and fruit/vegetable consumption. Additionally, support team member MVPA (via Fitbit) and secondary outcomes will be compared. We will also explore long-term MPVA and secondary outcomes in all groups at 6 months.

ELIGIBILITY:
Inclusion Criteria:

SURIVIVOR

* Diagnosed with early stage (I-II) endometrial cancer, any histology
* Received cancer care at Carilion Clinic after 1/1/2010
* At least 18 years of age
* Have adequate comprehension (reading and writing) of the English language
* Have a BMI ≥ 30 kg/m^2 at screening
* Have stable internet access or access to a smartphone with internet capabilities
* Meet the requirements of the Physical Activity Readiness Questionnaire(PARQ)
* Have the capacity to provide informed consent and are willing to provide informed consent
* SUPPORT TEAM--
* Were identified by a participant with endometrial cancer as a member of their support system
* Are at least 18 years of age
* Have adequate comprehension (reading and writing) of the English language
* Have stable internet access or access to a smartphone with internet capabilities
* Meet the requirements of the Physical Activity Readiness Questionnaire (PARQ)
* Have the capacity to provide informed consent and are willing to provide informed consent

Exclusion Criteria:

SURVIVOR

* Recurrent endometrial cancer
* Meeting physical activity guidelines set forth by the American Cancer Society at screening (greater than 150 minutes/week of moderate physical activity, or greater than 75 minutes/week of vigorous physical activity)
* SUPPORT TEAM: Have functional limitations requiring a walker, wheelchair, scooter, or other walking aid which limits their capacity to engage in the intervention safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Armbruster, MD MPH, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | FitEx-ECS | FitEx-ECS+ Yoga
Started | 18 | 35 | 58
Completed | 18 | 29 | 57
Not Completed | 0 | 6 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 1

BASELINE CHARACTERISTICS:
Population: Completion of all questions and survey information was not required for study enrollment. Data that was obtained is provided.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | FitEx-ECS | FitEx-ECS+ Yoga | Total
Number analyzed (Participants) | 18 | 29 | 57 | 104
Age, Continuous [Median (Full Range); unit: years] — Population: Not all participants included a date of birth so age could not be calculated
  years
    number analyzed (Participants) | 18 | 23 | 49 | 90
    (all) | 58 [39 to 77] | 55 [28 to 79] | 55.6 [20 to 87] | 55.5 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all enrolled participants completed all intake questionnaires.
  Participants
    number analyzed (Participants) | 18 | 22 | 47 | 87
    Female | 18 | 18 | 41 | 77
    Male | 0 | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all enrolled participants completed all intake questionnaires.
  Participants
    Hispanic or Latino | 0 | 0 | 1 | 1
    Not Hispanic or Latino | 18 | 20 | 48 | 86
    Unknown or Not Reported | 0 | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Not all enrolled participants completed all intake questionnaires. For the usual care group: a question about race was not included in the baseline survey unintentionally, therefore this information was not captured.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 23 | 47 | 70
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 18 | 6 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity of Endometrial Cancer Survivors
Description: Among survivors, compare changes in objective moderate-vigorous physical activity (MVPA) obtained from FitBits (continuous tracking) between intervention groups and usual care (FitEx-ECS vs. control and FitEx-ECS+yoga vs. control)
Time Frame: Change from baseline to 8 weeks (post-intervention)
Population: Minutes per day of moderate to vigorous physical activity (MVPA) over 7 days was compared from 8 weeks to baseline data. Participants need to have at least 4 days per week of wear time at each time point to be included.
Measure: Mean (Standard Deviation); unit: minutes per day of MVPA
Arm/Group | Usual Care | FitEx-ECS | FitEx-ECS+ Yoga
Number analyzed (Participants) | 16 | 8 | 14
minutes per day of MVPA | 3.7 (26.4) | 12.14 (40.75) | 3.15 (25.5)

2. Secondary Outcome: Quality of Life- Survivors
Description: Examine the change in quality of life (measured via Functional Assessment of Cancer Therapy - Endometrial (FACT-En)) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: physical well-being (0-28), social well-being (0-28), emotional well-being (0-28), functional well-being (0-28), endometrial cancer sub-scale (0-64); higher scores indicate better quality of life
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life Maintenance- Survivors
Description: Examine the change in quality of life (measured via Functional Assessment of Cancer Therapy - Endometrial) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: physical well-being (0-28), social well-being (0-28), emotional well-being (0-28), functional well-being (0-28), endometrial cancer sub-scale (0-64); higher scores indicate better quality of life
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

4. Secondary Outcome: Servings of Daily Fruits and Vegetables Maintenance- Survivors
Description: Examine the change in fruit/vegetable intake (measured via Behavioral Risk Factor Surveillance System (BRFSS F/V) survey) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

5. Secondary Outcome: Servings of Daily Fruits and Vegetables- Survivors
Description: as for outcome 4
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

6. Secondary Outcome: Flourishing- Survivors
Description: Examine the change in flourishing (measured via The Flourishing Index) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: 0-10, with higher scores indication more satisfaction/flourishing
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

7. Secondary Outcome: Flourishing Maintenance- Survivors
Description: as for outcome 6
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

8. Secondary Outcome: Yoga Self-Efficacy- Survivors
Description: Examine the change in yoga self-efficacy (measured via the Yoga Self-Efficacy Scale) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: (12-108) higher scores indicate higher efficacy for yoga
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

9. Secondary Outcome: Yoga Self-Efficacy Maintenance- Survivors
Description: as for outcome 8
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

10. Secondary Outcome: Social Support- Survivors
Description: Examine the change in social support (measured via the Sallis Social Support for Exercise Survey) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: higher numbers indicate more support
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

11. Secondary Outcome: Social Support Maintenance- Survivors
Description: as for outcome 10
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

12. Secondary Outcome: Self-compassion- Survivors
Description: Examine the change in self-compassion (measured via the Neff 12 item Self-Compassion Scale Short Form (SCS-SF) ) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: (1, 5) with higher scores indicating more self-compassion
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

13. Secondary Outcome: Self-compassion Maintenance- Survivors
Description: as for outcome 12
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

14. Secondary Outcome: Habit Formation- Survivors
Description: Examine the change in habit formation around exercise (measured via Self-Reported Behavior Automaticity Index) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring (1,7), higher scores indicate more automaticity/habit formation
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

15. Secondary Outcome: Habit Formation Maintenance- Survivors
Description: as for outcome 14
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

16. Secondary Outcome: Physical Activity Level (Active or Insufficiently Active) Maintenance- Survivors
Description: Examine the change in national physical activity goal attainment (measured via The Stanford Leisure-Time Activity Categorical Item (L-Cat)) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

17. Secondary Outcome: Physical Activity Level (Active or Insufficiently Active)- Survivors
Description: Examine the change in national physical activity goal attainment (measured via The Stanford Leisure-Time Activity Categorical Item (L-Cat)) between intervention and usual care conditions (FitEx-ECS versus control and FitEx-ECS+yoga versus control).
  Scoring: responses are categorical
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

18. Secondary Outcome: Moderate to Vigorous Physical Activity of Endometrial Cancer Survivors- Maintenance
Description: Among survivors, compare changes in objective moderate-vigorous physical activity (MVPA) obtained from FitBits between intervention groups and usual care (FitEx-ECS vs. control and FitEx-ECS+yoga vs. control)
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Moderate to Vigorous Physical Activity- Support Team Members
Description: Among survivors, compare changes in objective moderate-vigorous physical activity (MVPA) obtained from FitBits between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga)
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Moderate to Vigorous Physical Activity Maintenance- Support Team Members
Description: as for outcome 19
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Flourishing- Support Team Members
Description: Examine the change in flourishing (measured via The Flourishing Index) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga) Scoring: 0-10, with higher scores indication more satisfaction/flourishing
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Flourishing Maintenance- Support Team Members
Description: as for outcome 21
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Yoga Self-Efficacy- Support Team Members
Description: Examine the change in yoga self-efficacy (measured via the Yoga Self-Efficacy Scale) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga) Scoring: (12-108) higher scores indicate higher efficacy for yoga
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Yoga Self-Efficacy Maintenance- Support Team Members
Description: as for outcome 23
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Social Support- Support Team Members
Description: Examine the change in social support (measured via the Sallis Social Support for Exercise Survey) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga) Scoring: higher numbers indicate more support
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Social Support Maintenance- Support Team Members
Description: as for outcome 25
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Self-compassion- Support Team Members
Description: Examine the change in self-compassion (measured via the Neff 12 item Self-Compassion Scale Short Form (SCS-SF)) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga) Scoring: (1, 5) with higher scores indicating more self-compassion
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Self-compassion Maintenance- Support Team Members
Description: as for outcome 27
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Habit Formation- Support Team Members
Description: Examine the change in habit formation around exercise (measured via Self-Reported Behavior Automaticity Index) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga) Scoring (1,7), higher scores indicate more automaticity/habit formation
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Physical Activity Level (Active or Insufficiently Active)- Support Team Members
Description: Examine the change in national physical activity goal attainment (measured via The Stanford Leisure-Time Activity Categorical Item (L-Cat)) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga)
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Physical Activity Level (Active or Insufficiently Active) Maintenance- Support Team Members
Description: as for outcome 30
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Habit Formation Maintenance- Support Team Members
Description: as for outcome 29
Time Frame: Change from 8 weeks to 6 months (post-intervention)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Servings of Daily Fruits and Vegetables- Support Team Members
Description: Examine the change in fruit/vegetable intake (measured via Behavioral Risk Factor Surveillance System (BRFSS F/V) survey) between intervention groups (FitEx-ECS vs. FitEx-ECS+yoga)
Time Frame: Change from baseline to 8 weeks (post-intervention)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were observed for 10 weeks: one week at baseline, 8 weeks during the study, and one week 6 months after completing the intervention.
Arm/Group | Usual Care | FitEx-ECS | FitEx-ECS+ Yoga
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/29 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/57
Other Adverse Events (participants affected / at risk) | 0/18 | 0/29 | 0/57

LIMITATIONS AND CAVEATS:
Following randomization, 7 participants withdrew from participation due to changes in their ability to attend weekly meetings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT05737745/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT05737745/ICF_001.pdf